CLINICAL TRIAL: NCT04150952
Title: Physiological and Psychological Effects of Heart Rate Variability Based Training in Endurance Athletes
Brief Title: HRV-based Training Effects in Athletes
Acronym: HRV-btA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, María Carrasco Poyatos, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAL-HRV
Record Dates: First submitted 2019-10-24; First posted 2019-11-05 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Heart Rate Control; Athlete; Emotions
Keywords: Heart rate variability; Training; Endurance; Mood; Anxiety; Stress; maximal oxygen consumption
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRV-Group (Experimental): Athletes will train according to their basal HRV scores. If the resting HRV is higher tan their basal HRV, they will perform a high or moderate intensity training. If the resting HRV is lower, they will perform a low intensity training. If the resting HRV still lower, they will rest. They will not accumulate two or more days of high-moderate intensity training, nor two or more days of rest.
  Interventions: Other: HRV-based training
- TRAD-Group (Active Comparator): Athletes will train according to their trainer plan. Training will not be guided by their basal HRV scores.
  Interventions: Other: TRAD training

INTERVENTIONS:
Other: HRV-based training — Intervention based on HRV-guided training for the performance improvement of athletes. Pre-competitive HRV, subjective effort perception, anxiety and mood will also be analysed.
  Arms: HRV-Group
Other: TRAD training — Traditional endurance training
  Arms: TRAD-Group

SUMMARY:
Monitoring individual responses to training is an important key factor to prescribe to most effective training programs. Heart-rate variability (HRV) could be used for monitoring the training status of endurance athletes in order to detect the fatigue status and to assess the adaptation to training. This direct fatigue measuring method has been little used to prescribe or regulate exercise prescription. Moreover, it allows new possibilities for the training load prescription according to an athlete's status, the response to the training load, and the adaptation to training. Regardless HRV-guided training, the athlete performance could also be influenced by precompetitive mood and anxiety, which can also be reflected in the precompetitive HRV scores and the subjective effort perception.

DETAILED DESCRIPTION:
Monitoring individual responses to training is an important key factor to prescribe to most effective training programs. A promising variable that is able to reflect positive or negative training adaptation is cardiac autonomic regulation. In general, a decreased training status is associated with a lower power output at the same submaximal heart rate and a slower heart rate recovery, whereas an increased training status is associated with an increased power output, the same submaximal heart rate, and a faster heart rate recovery.

In this line, heart-rate variability (HRV), which focuses on the variability of successive R-R intervals, have gained popularity in monitoring the training status of endurance athletes. This tool enables the detection of fatigue status and assesses the adaptation to training. After high intensity training or a short-term overreached period, there is a decrease in the resting HRV values, reflecting the effect of the fatigue. In addition, the increase of the performance after a training period is related to an increase in resting HRV. This direct fatigue measuring method has been little used to prescribe or regulate exercise prescription. Moreover, this HRV-guided training, also called day-to-day periodization, allows new possibilities for the training load prescription according to an athlete's status, the response to the training load, and the adaptation to training.

On the other hand, regardless HRV-guided training, the athlete performance could also be influenced by precompetitive mood and anxiety, which can also be reflected in the precompetitive HRV scores and the subjective effort perception. This is another interesting line that pretends to be clarified in this study.

ELIGIBILITY:
Inclusion Criteria:

* Belonging to the Spanish Athletics Federation.
* Training and running in Spanish Athletics Federation contest during at least two years.
* Stay in the first third of the classification of the previous season last five races.

Exclusion Criteria:

* Cardiovascular pathologies.
* Parameters of blood pressure (BP) outside of normality.
* Respiratory problems diagnosed.
* Be in treatment of psychological problems.
* Regular consumption of drug (s) with direct or indirect effects on the Nervous System (e.g., anxiolytics, antidepressants, neuroleptics).
* Consumption of substances not permitted by the International Athletics Federation (IAF).
* Punctual consumption of medication that could alter the performance due to suffering some disease related to cardiorespiratory system (e.g., influenza).
* Do not attend at least the 90% of the workouts during the intervention.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-07 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
VO2max | Change from baseline VO2max at 8 weeks
  Maximal oxygen consumption in treadmill test

SECONDARY OUTCOMES:
maximal heart rate | Change from baseline maximal heart rate at 8 weeks
  maximal heart rate in the treadmill test
maximal speed | Change from baseline maximal speed at 8 weeks
  maximal speed in the treadmill test
ventilatory thresolds | Change from baseline ventilatory thresolds at 8 weeks
  ventilatory thresolds in the treadmill test
respiratory quotient | Change from baseline respiratory quotient at 8 weeks
  respiratory quotient in the treadmill test
Time in running test | Change from baseline time at 8 weeks
  Time in the 3000 meters running test
Lactate change | Change from baseline Lactate at 8 weeks
  Lactate change after the 3000m test
Speed in running test | Change from baseline speed at 8 weeks
  Speed in the 3000 meters running test
Heart rate in running test | Change from baseline heart rate at 8 weeks
  Heart rate in the 3000 meters running test
Börg scale after running test | Through study completion (8 weeks)
  Subjective perceived exertion. Scores goes from 0 to 10. Higher scores indicate a higher perceived exertion.
LnrMSSD score | Through study completion (8 weeks)
  Parasympathetic tone and recovery indicator. There are no minimum or maximum values. They depend on the athlete recovery state. Higher scores indicate a better outcome.
Mood score | Through study completion (8 weeks)
  Precompetitive mood levels. Instrument: Profile of Mood States. Scores goes from 0 (low mood) to 4 (high mood).
Anxiety score | Through study completion (8 weeks)
  Precompetitive anxiety levels. Instrument: Revised Competitive State Anxiety Inventory-2. Scores goes from 1 (no anxiety) to 4 (a lot of anxiety).

OTHER OUTCOMES:
Fat mass | Change from baseline body composition at 8 weeks
  Percentage of fat mass
Muscle mass | Change from baseline body composition at 8 weeks
  Percentage of muscle mass
Bone mass | Change from baseline body composition at 8 weeks
  Percentage of bone mass
Body water | Change from baseline body composition at 8 weeks
  Percentage of body water
Height | Change from baseline height at 8 weeks
  Height in meters
Weight | Change from baseline weight at 8 weeks
  Weight in kilograms
Heart Rate Variability Change (LnrMSSD) | Change from Baseline Heart Rate Variability at 8 weeks
  Parasympathetic tone and recovery indicator

CONTACTS AND LOCATIONS:
Overall Officials: Alberto González Quílez, Master, Study Chair — Universidad de Almeria; Antonio Granero-Gallegos, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- University of Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: No